CLINICAL TRIAL: NCT01733121
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Titration Study to Assess the Safety, Tolerability, and Efficacy of NBI-98854 for the Treatment of Tardive Dyskinesia
Brief Title: NBI-98854 Dose Titration Study for the Treatment of Tardive Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-1202
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBI-98854 (Experimental): Dose titration to determine a subject's optimal dose in the range of 25 to 75 mg NBI-98854. Dose titration is performed in increments of 25 mg. NBI-98854 administered as one (1) 25 mg capsule, two (2) 25 mg capsules, or one (1) 25 mg capsule and one (1) 50 mg capsule by mouth, taken every morning between 7:00am - 10:00am for 6 weeks.
  Interventions: Drug: NBI-98854
- Placebo (Placebo Comparator): Capsule containing no active substance, manufactured to mimic NBI-98854 25 mg and 50 mg capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-98854 — 25 mg capsule
  Arms: NBI-98854
Drug: NBI-98854 — 50 mg capsule
  Arms: NBI-98854
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of NBI-98854 (titrated to a subject's optimal dose in the range of 25 to 75 mg) administered once daily for the treatment of Tardive Dyskinesia (TD) symptoms.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, dose-titration study to evaluate the efficacy, safety, and tolerability of NBI-98854 (titrated to subject's optimal dose in the range of 25 to 75 mg) compared to placebo, administered once daily (q.d.) for a total of 6 weeks of treatment. Approximately 90 medically stable male and female subjects with one of the following clinical diagnoses will be enrolled: schizophrenia or schizoaffective disorder with neuroleptic-induced TD; mood disorder with neuroleptic-induced TD; or gastrointestinal disorder with metoclopramide-induced TD.

For subjects randomized to active treatment, the starting dose will be 25 mg NBI 98854, which may be escalated in increments of 25 mg every 2 weeks to a maximum of 75 mg to achieve an optimal dose of NBI-98854 for each subject

ELIGIBILITY:
Inclusion Criteria:

* Have one of the following clinical diagnoses for at least 3 months prior to screening a) schizophrenia or schizoaffective disorder; b) mood disorder; or c) gastrointestinal disorder (e.g., gastroparesis, gastroesophageal reflux disease)
* Have a clinical diagnosis of neuroleptic-induced tardive dyskinesia for at least 3 months prior to screening.
* Be receiving a stable dose of antipsychotic medication for a minimum of 30 days before study start. Subjects who are not using antipsychotic medication must have stable psychiatric status.
* Have the doses of concurrent medications and the conditions being treated be stable for a minimum of 30 days before study start and be expected to remain stable during the study.
* Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal birth control during the study.
* Female subjects must not be pregnant.
* Be in good general health and expected to complete the clinical study as designed.
* Have a body mass index (BMI) of 18 to 38 kg/m2 (both inclusive).
* Have a negative urine drug screen (negative for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, opiates, or cannabinoids) at screening and study start, except for any subject receiving a stable dose of benzodiazepine.
* Have a negative alcohol breath test at screening and study start.

Exclusion Criteria:

* Have an active clinically significant unstable medical condition within 1 month (30 days) prior to screening.
* Have a history of substance dependence or substance (drug) or alcohol abuse within the 3 months before study start(nicotine and caffeine dependence are not exclusionary).
* Have a known history of neuroleptic malignant syndrome.
* Have a significant risk of suicidal or violent behavior.
* Receiving any excluded concomitant medication such as reserpine, metoclopramide, stimulants, or tetrabenazine.
* Receiving medication for the treatment of tardive dyskinesia.
* Have a positive human immunodeficiency virus antibody, (HIV-Ab), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody result at screening or have a history of positive result.
* Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study.
* Have an allergy, hypersensitivity, or intolerance to tetrabenazine.
* Have had previous exposure with NBI-98854.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD, Study Director — Neurocrine Biosciences
Locations (21):
- United States (20):
  - Costa Mesa, California
  - Fountain Valley, California
  - Oceanside, California
  - Englewood, Colorado
  - Boca Raton, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - Farmington Hills, Michigan
  - Beachwood, Ohio
  - Middleburg Heights, Ohio
  - Conshohocken, Pennsylvania
  - Phoenixville, Pennsylvania
  - Bedford, Texas
  - DeSoto, Texas
  - Houston, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Richland, Washington
- Caguas, Puerto Rico

REFERENCES:
- [Derived] Sajatovic M, Alexopoulos GS, Burke J, Farahmand K, Siegert S. The effects of valbenazine on tardive dyskinesia in older and younger patients. Int J Geriatr Psychiatry. 2020 Jan;35(1):69-79. doi: 10.1002/gps.5218. Epub 2019 Oct 31. PMID 31617235
- [Derived] Grigoriadis DE, Smith E, Hoare SRJ, Madan A, Bozigian H. Pharmacologic Characterization of Valbenazine (NBI-98854) and Its Metabolites. J Pharmacol Exp Ther. 2017 Jun;361(3):454-461. doi: 10.1124/jpet.116.239160. Epub 2017 Apr 12. PMID 28404690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with schizophrenia or schizoaffective disorder with tardive dyskinesia (TD), a mood disorder with TD, or a GI disorder with TD from 29 centers in the United States and Puerto Rico. The last patient completed in December 2013.
Groups:
- Placebo: Participants received Placebo capsule (matching valbenazine capsules) once daily for 6 weeks.
- Valbenazine: Participants could receive valbenazine 25mg once daily for 2 weeks, then 50mg once daily for 2 weeks, then 75mg once daily for 2 weeks (a total of 6 weeks); flexible dose escalation.
Period: Double-Blind Period (Week 0 to 6)
Arm/Group | Placebo | Valbenazine
Started | 51 | 51
Completed | 44 | 46
Not Completed | 7 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Non-compliance | 3 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Period: Follow-Up Period (Week 6 to 8)
Arm/Group | Placebo | Valbenazine
Started | 44 | 46
Completed | 44 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (all randomized subjects who received at least one dose of study drug).
Groups:
- Placebo: Participants received Placebo capsule (matching valbenazine capsules) daily for 6 weeks.
- Valbenazine: Participants received valbenazine 25mg once daily for 2 weeks, then 50mg once daily for 2 weeks, then 75mg once daily for 2 weeks (a total of 6 weeks).
- Total: Total of all reporting groups
Arm/Group | Placebo | Valbenazine | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Full Range); unit: years] | 55.6 [34 to 78] | 56.7 [32 to 78] | 56.2 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 27 | 30 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska native | 1 | 0 | 1
  American Indian/Alaska native, Caucasian | 1 | 0 | 1
  Black/African American | 16 | 18 | 34
  Caucasian | 30 | 33 | 63
  Other/mixed | 1 | 0 | 1
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28.19 [18.0 to 38.3] | 29.02 [18.1 to 42.0] | 28.62 [18.0 to 42.0]
Disease Category [Count of Participants; unit: Participants]
  Schizophrenia or schizoaffective disorder | 30 | 28 | 58
  Mood disorder | 18 | 20 | 38
  Gastrointestinal disorder | 1 | 3 | 4
Age at TD Diagnosis [Mean (Full Range); unit: years] — Population: Date of diagnosis was not available for some subjects.
  years
    number analyzed (Participants) | 36 | 39 | 75
    (all) | 49.5 [23 to 77] | 48.9 [25 to 70] | 49.2 [23 to 77]
BPRS Total Score [Mean (Full Range); unit: units on a scale] — The Brief Psychiatric Rating Scale (BPRS) is a clinician-rated tool designed to assess change in the severity of psychopathology in patients with schizophrenia and other psychotic disorders (Overall and Gorham, 1962, 1988). The severity of each of the 18 items of the BPRS is rated on a scale of 1 (not present) to 7 (extremely severe) (total score range: 18 to 126). Higher scores represent greater symptom severity.
  units on a scale | 30.1 [19 to 49] | 30.1 [19 to 48] | 30.1 [19 to 49]
Baseline AIMS Total Dyskinesia Score [Mean (Standard Deviation); unit: units on a scale] — The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity. Population: Includes subjects with a central video raters' AIMS dyskinesia total score change from baseline value at Week 6
  units on a scale
    number analyzed (Participants) | 44 | 45 | 89
    (all) | 7.9 (4.5) | 8.0 (3.5) | 8.0 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score Change From Baseline at Week 6
Description: The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.
Time Frame: Baseline and Week 6
Population: Per protocol analysis set (subjects in the ITT analysis set that had an evaluable, blinded, central video raters' AIMS dyskinesia total score change from baseline value at Week 6, had a quantifiable NBI-98782 plasma concentration at Week 6 [for subjects in the NBI-98854 group], and had no efficacy-related important protocol deviations)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Valbenazine: Participants first received valbenazine 25mg once daily for 2 weeks, then 50mg once daily for 2 weeks, then 75mg once daily for 2 weeks (a total of 6 weeks).
Arm/Group | Placebo | Valbenazine
Number analyzed (Participants) | 44 | 32
units on a scale | -0.3 (1.1) | -3.4 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Valbenazine; Test type: Other; p < .0001, ANCOVA; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-4.5 to -1.6], Standard Error of Mean 0.7

2. Secondary Outcome: Clinical Global Impression - Global Improvement of TD (CGI-TD) at Week 6
Description: Clinician's perspective of the participant's overall improvement of TD symptoms over time. The CGI-TD is based on a 7-point scale (range: 1=very much improved to 7=very much worse).
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Valbenazine
Number analyzed (Participants) | 44 | 32
units on a scale | 3.1 [2.5 to 3.6] | 2.2 [1.6 to 2.9]
Statistical Analysis 1: Comparison: Placebo vs Valbenazine; Test type: Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.2 to -0.4], Standard Error of Mean 0.2

3. Secondary Outcome: AIMS Dyskinesia Total Score Change From Baseline at Week 6
Description: as for outcome 1
Time Frame: Week 6
Population: Intent to Treat (ITT) analysis set (all subjects in the safety analysis set with an evaluable, blinded, central video raters' AIMS dyskinesia total score change from baseline value at one or more scheduled assessment times during the double-blind treatment period)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Placebo: Participants received Placebo capsule (matching NBI-98854 capsules) once daily for 6 weeks.
- NBI-98854: Participants first received NBI-98854 25mg once daily for 2 weeks, then 50mg once daily for 2 weeks, then 75mg once daily for 2 weeks (a total of 6 weeks).
Arm/Group | Placebo | NBI-98854
Number analyzed (Participants) | 44 | 45
units on a scale | -0.2 [-2.4 to 2.0] | -2.6 [-4.9 to -0.3]
Statistical Analysis 1: Comparison: Placebo vs NBI-98854; Test type: Other; p = 0.0005, ANCOVA; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-3.7 to -1.1], Standard Error of Mean 0.7

4. Secondary Outcome: Clinical Global Impression - Global Improvement of TD (CGI-TD) at Week 6
Description: as for outcome 2
Time Frame: Week 6
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Valbenazine
Number analyzed (Participants) | 44 | 45
units on a scale | 3.1 [2.5 to 3.6] | 2.2 [1.7 to 2.8]
Statistical Analysis 1: Comparison: Placebo vs Valbenazine; Test type: Other; p < .0001, ANOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.2 to -0.5], Standard Error of Mean 0.2

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Groups:
- Placebo: Participants received Placebo capsule (matching valbenazine capsules) daily for 6 weeks followed by 2 weeks posttreatment period.
- Valbenazine: Participants first received valbenazine 5mg once daily for 2 weeks, then 50mg once daily for 2 weeks, then 75mg once daily for 2 weeks (a total of 6 weeks) followed by 2 weeks posttreatment period.
Arm/Group | Placebo | Valbenazine
All-Cause Mortality (participants affected / at risk) | 1/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 2/49 | 0/51
Other Adverse Events (participants affected / at risk) | 11/49 | 16/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Valbenazine (N=51)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Valbenazine (N=51)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 5 (5)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.